CLINICAL TRIAL: NCT05561361
Title: The Effect of Selective Adrenal Artery Embolism on Vascular Endothelial Function in Patients With Primary Aldosteronism Based on Brachial Artery Flow-mediated Relaxation
Brief Title: The Effect of SAAE on Vascular Endothelial Function in PA Patients
Status: Recruiting | Type: Observational
Sponsor: Second Affiliated Hospital of Nanchang University (Other)
Responsible Party: Sponsor
Other Study IDs: IIT-O-2021-032
Record Dates: First submitted 2022-09-27; First posted 2022-09-30 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-05

CONDITIONS: Primary Aldosteronism
Keywords: primary aldosteronism; selective adrenal artery embolization; vascular endothelial function
MeSH Terms: conditions — Hyperaldosteronism | interventions — Spironolactone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SAAE group: Subjects received super selective adrenal artery embolization treatment
  Interventions: Procedure: Super selective adrenal artery embolization
- Spironolactone group: Subjects received spironolactone treatment
  Interventions: Drug: Spironolactone

INTERVENTIONS:
Procedure: Super selective adrenal artery embolization — Superselective adrenal arterial embolization is an operation to inject embolic agent into adrenal artery through catheter to embolize part of adrenal gland, so as to reduce the secretion of adrenal hormone and reduce blood pressure.
  Other Names: SAAE
  Groups: SAAE group
Drug: Spironolactone — Aldosterone receptor antagonists are recommended by guidelines for the treatment of bilateral primary aldosteronism.
  Groups: Spironolactone group

SUMMARY:
The study aims to assess the effect of superselective adrenal arterial embolization on vascular endothelial function in patients with primary aldosteronism based on brachial artery flow-mediated relaxation

DETAILED DESCRIPTION:
After being informed about the study and potential risks,all patients giving written informed consent will undergo a 2-week screening period to determine eligibility for study entry.At week 0,patients who meet the eligibility requirements will be divided into Superselective adrenal arterial embolization group or spironolactone therapy group,according to the patient's surgical indications and wishes.

ELIGIBILITY:
Inclusion Criteria:

* (1)Aged 18-75 years, males and females;
* (2)Blood pressure ≥ 140/90 mmHg on at least three non-same-day office visits without antihypertensive medication or 24-hour ambulatory blood pressure averaging >130/80 mmHg throughout the day or averaging >135/85 mmHg during the day;
* (3)Primary aldosteronism was diagnosed in accordance with the 2016 international society of Endocrinology clinical guidelines after strict drug elution;
* (4)Contraindications to spironolactone-free administration;
* (5)No surgical intention or surgical contraindications, and willing to accept drug treatment or percutaneous superselective adrenal artery embolization;
* (6)The anatomy of adrenal arteriography is suitable for selective adrenal artery embolization.

Exclusion Criteria:

* (1)Secondary hypertension of other causes;
* (2)Pregnant women or those who have a fertility plan in the next year;
* (3)Glomerular filtration rate EGFR < 45 ml/min/1.73m^2;
* (4)History of severe contrast allergy;
* (5)Hyperkalemia;
* (6)Patients with other serious organic diseases or life expectancy < 12 months can not tolerate the treatment of super selective adrenal artery embolizatio;
* (7)The diameter of adrenal space occupying lesions was more than 2 cm;
* (8)A history of myocardial infarction, syncope, cerebral hemorrhage or cerebral infarction within 3 months before the informed consent;
* (9)The results of this study will be affected during the period when patients are enrolled or will participate in other clinical studies.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who were diagnosed with primary aldosteronism and underwent adrenal vein sampling at the Second Affiliated Hospital of Nanchang University.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
endothelial function | 1 month after SAAE
  Brachial artery endothelial function measured by flow-mediated dilation(FMD)
endothelial function | 12 months after SAAE
  Brachial artery endothelial function measured by flow-mediated dilation(FMD)

SECONDARY OUTCOMES:
PAC | 1 month after SAAE
  plasma aldosterone concentration
PAC | 12 months after SAAE
  plasma aldosterone concentration
PRA | 1 month after SAAE
  plasma renin activity
PRA | 12 months after SAAE
  plasma renin activity
ARR | 1 month after SAAE
  aldosterone-to-renin ratio
ARR | 12 months after SAAE
  aldosterone-to-renin ratio
Serum potassium | 1 month after SAAE
  Serum potassium
Serum potassium | 12 months after SAAE
  Serum potassium
serum creatinine | 1 month after SAAE
  serum creatinine
serum creatinine | 12 months after SAAE
  serum creatinine

CONTACTS AND LOCATIONS:
Overall Officials: Yifei Dong, Study Director — Second Affiliated Hospital of Nanchang University
Locations (1):
- The Second Affiliated Hospital of Nanchang University, Nanchang, China